CLINICAL TRIAL: NCT00103805
Title: Improved Language Acquisition With Levodopa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KS-LD_01
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: language acquisition; plasticity; stroke recovery; associative learning
MeSH Terms: interventions — Levodopa

INTERVENTIONS:
Drug: levodopa

SUMMARY:
The purpose of this study is to determine whether the non-daily administration of levodopa is effective in boosting semantic language acquisition in healthy subjects.

DETAILED DESCRIPTION:
Our prior work using a between-subject design shows that daily administration of d-amphetamine or the dopamine precursor levodopa over the course of five days markedly improves word learning success in healthy subjects. In this randomized, placebo-controlled, double-blind clinical trial, we probe whether the effect can be replicated using a within-subject design, with administration of levodopa and placebo on alternate days for a total period of 10 days.

The expected scientific results will strengthen the basis for transferring neuromodulatory interventions from the laboratory to stroke patients with language dysfunctions. Because of the heterogeneity of stroke patients, only a within-subject design can be used to probe the effects of pharmacological adjuncts to language therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* 20-35 years old
* Right handedness

Exclusion Criteria:

* Neurological/psychiatric/metabolic/cardiac disorders
* Asthma
* Known allergic reactions to one of the experimental drugs
* Other drugs affecting the central nervous system
* Leisure drug ingestion during the past 4 weeks (urine test)
* Smoking cessation during the past 2 weeks
* > 6 cups of coffee or energy drinks per day
* > 10 cigarettes per day
* > 50 grams of alcohol per day

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2003-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Boost in language learning success through levodopa compared to placebo

SECONDARY OUTCOMES:
Stability of language learning success after one month

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Breitenstein, PhD, Study Director — Dept. of Neurology, University of Muenster, Germany; Stefan Knecht, MD, Study Chair — Dept. of Neurology, University of Muenster, Germany
Locations (1):
- Dept. of Neurology, University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Breitenstein C, Wailke S, Bushuven S, Kamping S, Zwitserlood P, Ringelstein EB, Knecht S. D-amphetamine boosts language learning independent of its cardiovascular and motor arousing effects. Neuropsychopharmacology. 2004 Sep;29(9):1704-14. doi: 10.1038/sj.npp.1300464. PMID 15114342